CLINICAL TRIAL: NCT01257035
Title: The Predictive Value of 18F-FAZA-PET/CT in Neoadjuvant Radiation for Patients With Locally Advanced Rectum Cancer
Brief Title: Predictive Value of 18F-FAZA in Rectum Cancer
Acronym: FAZA
Status: Terminated | Type: Observational
Why Stopped: The logistics of this trial (incl. supply of tracer) in connection with the patients' treatment course caused the inclusion rate to be very slow.
Sponsor: Vejle Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S-20100054
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Locally Advanced Rectum Cancer
Keywords: Rectum cancer; FAZA; 18F-FAZA-PET/CT; Radiotherapy; Chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 18F-FAZA-PET/CT
  Interventions: Other: 18F-FAZA-PET/CT

INTERVENTIONS:
Other: 18F-FAZA-PET/CT — Contrast fluid injected prior to scan

SUMMARY:
The primary purpose of the study is to investigate 18F-FAZA-PETs role as predictor of response to neoadjuvant chemoradiation of locally advanced rectum cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histopatologically verified adenocarcinoma in the rectum
* T4 tumor eller T3 tumor < 10 cm from the anus and < 5 mm from the mesorectal fascie measured by MR scan. At the distal part of the rectum the distance to the mesorectal fascie is < 5 mm and therefore all T3 tumors are included in this area
* Suitable for preoperative radiation and chemotherapy
* No distant metastases
* Age >18 years
* Hematology ANC ≥1.5x10^9/l. Thrombocytes ≥ 100x10^9/l.
* Biochemistry Bilirubin ≤ 3 x UNL. ALAT ≤ 5 x UNL
* Creatinine ≤ UNL
* Contraception for fertile women
* Written and orally informed consent

Exclusion Criteria:

* Other malignant disease within 5 years, excl. non-melanotic skin cancer
* Previous radiation treatment of the pelvis
* Pregnant or breastfeeding women
* Surgery within 6 weeks prior to enrollment
* Serious concurrent medical disease
* Enrollment in study "A prospective observational study of patients with rectum cancer after concomitant radiation and chemotherapy", where the patients are potientially not operated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectum cancer receiving preoperative radiation treatment and concomitant chemotherapy at the Dept. of Oncology, Vejle Hospital.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Response to chemoradiotherapy measured by TRG | 8 weeks after chemoradiation treatment

SECONDARY OUTCOMES:
Recurrence free survival | From date of inclusion till date of verified recurrence
Survival | From date of inclusion till date of death by any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Vejle Hospital, Vejle, Denmark